CLINICAL TRIAL: NCT02044315
Title: Prevention of Inappropriate ICD Shocks
Acronym: RISSY-ICD
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Yuksek Ihtisas Hospital (Other)
Responsible Party: Principal Investigator, Serkan Cay, Associate Professor, Yuksek Ihtisas Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: SNY-168
Record Dates: First submitted 2014-01-21; First posted 2014-01-23 (Estimated); Last update posted 2014-01-23 (Estimated); Status verified 2014-01

CONDITIONS: Inappropriate ICD Therapy; Appropriate ICD Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conventional (Sham Comparator): Conventional ICD programming
  Interventions: Device: ICD programming
- High-zone (Experimental): High-zone ICD programming
  Interventions: Device: ICD programming

INTERVENTIONS:
Device: ICD programming

SUMMARY:
The aim of the present study is to investigate whether increasing detection zones can effectively reduce inappropriate ICD therapies in primary prevention patients.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years
* Cardiomyopathy (ischemic or not)
* Current accepted indication for ICD implantation

Exclusion Criteria:

* Previous device implantation
* Secondary prevention patients
* Pregnancy,
* Primary electrical disorders,
* Patient refusal,
* <1 year of expected mortality

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2012-01; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
First total inappropriate therapy | 12 months
  Occurence of first total inappropriate therapy at 12-month follow-up
Occurence of first total appropriate therapy at 12-month follow-up | 12 months
  Occurence of first total appropriate therapy at 12-month follow-up

SECONDARY OUTCOMES:
All-cause mortality | 12 months
  Occurence of all-cause mortality at 12-month follow-up
Hospitalization for heart failure | 12 months
  Occurence of hospitalization for heart failure at 12-month follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Yuksek Ihtisas Hospital, Ankara, Cankaya, Turkey (Türkiye)